CLINICAL TRIAL: NCT00004351
Title: Study of Phenotype and Genotype Correlations in Patients With Contiguous Gene Deletion Syndromes
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Collaborators: Baylor College of Medicine (Other)
Organization: Office of Rare Diseases (ORD) (NIH)
Other Study IDs: 199/11914; BCM-H4299
Record Dates: First submitted 1999-10-18; First posted 1999-10-19 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2003-10

CONDITIONS: Williams Syndrome; Angelman Syndrome; Prader-Willi Syndrome; Shprintzen Syndrome; Smith-Magenis Syndrome; DiGeorge Syndrome; Chromosome Abnormalities
Keywords: Angelman syndrome; DiGeorge syndrome; Prader-Willi syndrome; Shprintzen syndrome; Smith-Magenis syndrome; Williams syndrome; genetic diseases and dysmorphic syndromes; neurologic and psychiatric disorders; rare disease
MeSH Terms: conditions — Williams Syndrome; Angelman Syndrome; Prader-Willi Syndrome; DiGeorge Syndrome; Smith-Magenis Syndrome; Chromosome Aberrations; Genetic Diseases, Inborn; Neurologic Manifestations; Mental Disorders; Rare Diseases

SUMMARY:
OBJECTIVES: I. Investigate phenotype and genotype correlations in patients with Smith-Magenis syndrome (SMS) associated with del(17p11.2).

II. Clinically evaluate SMS patients with unusual deletions or duplication of proximal 17p.

III. Clinically evaluate patients with Williams syndrome with molecular characterization of 7q11.23.

IV. Perform clinical studies of Prader-Willi, Angelman, DiGeorge, and Shprintzen syndrome patients with unique molecular findings in 15q11q13 or 22q11.2.

V. Perform genotype and phenotype correlations in Prader-Willi patients, particularly those with loss of expression of only some of the imprinted transcripts in 15q11-q13.

VI. Evaluate putative Angelman syndrome patients who do not have classic large deletion, uniparental disomy, or imprinting mutations, and perform molecular studies of the Angelman gene, UBE3A, and identify mutations of this gene.

VII. Investigate phenotype and genotype correlations in patients with terminal deletions of chromosome 1p.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: Patients undergo clinical, cytogenetic, and molecular studies. These include radiographic, neurologic, developmental, and 24 hour sleep studies, ophthalmologic, otolaryngologic, speech and language, and audiologic exams, echocardiogram, and renal ultrasound.

Smith-Magenis patients are also evaluated with the following: urine melatonin levels during day and night hours; anthropometrics; sleep and behavioral history; and renal, immunologic, and cholesterol studies. A clinical and phenotypic map is constructed.

When appropriate, parental chromosome analysis is performed.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics-- Contiguous gene deletion syndrome, e.g.: Smith-Magenis syndrome Williams syndrome DiGeorge syndrome Shprintzen syndrome (velo-cardio-facial syndrome) Prader-Willi syndrome Angelman syndrome Deletion of chromosome 1p Patient age: Any age

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20
Dates: Start 1999-09

CONTACTS AND LOCATIONS:
Overall Officials: James R. Lupski, Study Chair — Baylor College of Medicine
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States